CLINICAL TRIAL: NCT03143075
Title: Do Omega-3 Fatty Acids Have an Antidepressant Effect in Patients With Signs of Peripheral Inflammation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017150
Record Dates: First submitted 2017-04-20; First posted 2017-05-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Match/mismatch design (based on CRP levels), all subjects receive the same dose of EPA, no one receives placebo. Raters are blind to "Inflammation group" or "Non-inflammation group" allocation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Raters are blind to "Inflammation group" or "Non-inflammation group" allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inflammation group (Active Comparator): Subjects with CRP≥3, will receive eicosapentaenoic acid enriched omega-3 fatty acids, 2 g/day, for 8 weeks, added to their pre-stabilized antidepressant medication
  Interventions: Dietary Supplement: Eicosapentaenoic acid enriched omega-3 fatty acids, 2 g/day
- Non-inflammation group (Active Comparator): Subjects with CRP<3, will receive eicosapentaenoic acid enriched omega-3 fatty acids, 2 g/day, for 8 weeks, added to their pre-stabilized antidepressant medication
  Interventions: Dietary Supplement: Eicosapentaenoic acid enriched omega-3 fatty acids, 2 g/day

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic acid enriched omega-3 fatty acids, 2 g/day — Eicosapentaenoic acid enriched omega-3 fatty acids, 2 g/day, added to pre-stabilized antidepressant medication

SUMMARY:
In this study, the investigators will stratify depressed subjects a priori based on CRP levels to test the hypothesis that eicosapentaenoic (EPA) would be more efficacious to treat depression in subjects with high CRP levels compared to subjects with low CRP levels.

Depressed subjects, with ongoing stabilized antidepressive treatment who remain clinically depressed, will be enrolled in an "Inflammation group" or in a "Non-inflammation group" depending on baseline levels of CRP. Subjects in both groups will receive EPA enriched omega-3 fatty acids for 8 weeks, added to their pre-stabilized antidepressant medication.

DETAILED DESCRIPTION:
Background

Increased mean levels of peripheral inflammatory markers have repeatedly been reported in individuals with major depression compared to controls, although there is considerable overlap between groups. As further evidence for a role of inflammation in major depression, 20-60% of patients receiving treatment for viral hepatitis and certain forms of cancer with the cytokine interferon-alpha will develop depressive symptoms. Interestingly, some authors have suggested that the association between inflammation and depression is symptom specific, i.e. there might be a subtype of "inflammation-related depression" with a specific phenotype. Although it still remains unclear if the immune abnormalities often seen in depressed subjects derive from changes in the periphery or in the central nervous system (or both), animal studies have shown that by counteracting the effects of pro-inflammatory cytokines in either the blood or the brain, depressive-like behavior in animals can be mitigated. These animal studies, along with data from several clinical studies pertaining to this, suggest that interventions primarily targeting peripheral inflammation may be useful in treating psychiatric symptoms. Although the exact mechanisms by which increased inflammation may give rise to depressive symptoms remain unclear, there are several potential downstream pathways that may be involved including accelerated cellular aging, mitochondrial dysfunction, and oxidative stress.

In search for a potential antidepressant that could be tested in clinical trials in which subjects are selected a priori based on inflammatory markers, the investigators turn to eicosapentaenoic (EPA), an omega-3 (n-3) fatty acid with anti-inflammatory properties. The ability of dietary n-3 fatty acids to mitigate the inflammatory response has been shown in human and animal studies. EPA and Docosahexaenoic acid (DHA) are the two major n-3 fatty acids found in oily fish and fish oil supplements, and both have shown anti-inflammatory properties. Supplementation of EPA and DHA in individuals with cardiovascular disease results in decreased plasma levels of CRP. N-3 fatty acids also have several other anti-inflammatory properties including i) Decreased chemotaxis of neutrophils and monocytes, ii) Decreased expression of adhesion molecules (e.g. ICAM & VCAM) on the surface of immune cells and in the circulation, iii) Decreased production of prostaglandins, iv) Increased synthesis of anti-inflammatory molecules such as resolvins and protectins, and v) Inhibition of T-cell proliferation. The mechanisms underlying these effects are not fully understood but likely involves n-3 fatty acids acting via cell surface and intracellular receptors controlling inflammatory cell signaling and gene expression patterns. In addition to the well-established anti-inflammatory effects of n-3 fatty acids, they may also have beneficial effects on oxidative stress and cell aging parameters such as leukocyte telomere length and telomerase activity. However, more research is needed in order to confirm these relationships, and therefore the investigators will, in addition to assessing inflammatory markers, also study the effects of n-3 fatty acids on markers of cellular aging and oxidative stress.

Some, but not all, previous studies have shown that EPA is superior to placebo in treating unipolar or bipolar depression. Several caveats have, however, been issued when interpreting the results from these studies, including small and perhaps clinically irrelevant effect sizes, as well as potential publication bias. Generally, n-3 preparations with high doses of EPA relative to DHA have been shown to be more efficacious in treating depression. Interestingly, a double blind placebo-controlled RCT showed that that EPA (but not DHA) was effective in preventing interferon-alpha induced depression in hepatitis C subjects, consistent with the notion that EPA may have antidepressant effect in "inflammatory depression". In line with this notion, a recent a proof-of-concept study showed that high inflammation at baseline was associated with a better antidepressant effect of EPA, but not DHA, enriched n-3 compared to placebo. That study stratified subjects post-hoc based on inflammatory markers, whereas our approach will be to select study subjects a priori based on validated cut-offs for CRP. This is the next step in developing a personalized medicine paradigm for depression.

The main aims of the study are to test if i) EPA enriched n-3 (added to stabilized ongoing treatment) is efficacious in treating depressed patients, but only in subjects with prospectively ascertained elevations in baseline CRP, ii) Changes in inflammatory markers over the course of treatment mediate this effect, and iii) Clinical trial designs utilizing prospectively-ascertained biomarkers to predict response are feasible and thereby pave the way for personalized medicine in psychiatry.

Specific objective 1: To determine whether the antidepressant effect of n-3 EPA is greater in the Inflammation group than in the Non-inflammation group, controlling for baseline depression rating.

Hypothesis (H) 1: The antidepressant effect of n-3 EPA is greater in the Inflammation group than in the Non-inflammation group.

Specific objective 2: To determine whether changes in inflammatory, oxidative stress and cell aging markers from baseline to end of treatment correlate with antidepressant effect.

H 2: Change in inflammatory and cell aging markers with n-3 EPA treatment will be directly correlated with changes in depression ratings.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female, aged 18-80.
2. Fulfilling the DSM criteria for a current depressive episode, unipolar (symptom duration> 4 weeks) as determined by the study physician
3. HAM-D-17 score ≥ 15 (Rapaport, Nierenberg et al. 2016)
4. A Clinical Global Impression Severity Score ≥ 3 (Rapaport, Nierenberg et al. 2016)
5. All subjects should be stable on antidepressants or mood stabilizers ≥6 weeks.
6. Willing to not significantly modify their diet from the time they sign consent through the end of study participation.

Exclusion Criteria:

1. Serious or unstable medical illness that in the investigator's opinion could compromise response to treatment or interpretation of study results. Examples: Malignancy not in remission for at least 1 year, Active autoimmune disorder or inflammatory bowel disease, Insulin-dependent diabetes mellitus.
2. Known or suspected allergy to the study compounds.
3. Ongoing infection.
4. Ongoing pregnancy or breast-feeding
5. A diagnosis of psychotic disorder, bipolar disorder, mental retardation dementia, or individual whom, due to other causes, lack the ability to make an informed decision.
6. Ongoing ECT.
7. Concomitant use of anticoagulants or known bleeding disorder.
8. Patients who, in the investigator's judgment, pose a current, serious suicidal or homicidal risk.
9. A diagnosis for any Substance Use Disorder (except nicotine or caffeine) in the 3 months prior to the screening visit.
10. Any medications (within 1 week of baseline or during the trial) that might confound the biomarker findings, including: Regular ingestion of NSAIDs or COX-2 inhibitors, or any use of oral steroids, immunosuppressants, interferon, chemotherapy (Patients will be instructed not to take an NSAID, COX-2 inhibitor or Aspirin in the 24 hours prior to a biomarker assessment visit).
11. Patients who have taken supplements with omega-3 fatty acids for more than three consecutive days in the preceding month.
12. Within 4 weeks of starting psychotherapy or planning to start psychotherapy during the study
13. Active participation in other clinical studies with ongoing study visits

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | 8 weeks
  Absolute difference between baseline and week 8 of the total sum of the HAM-D-17

SECONDARY OUTCOMES:
Response | 8 weeks
  Clinical "response" is defined as a 50% or greater reduction in depressive symptoms after treatment.
Change in depressed mood | 8 weeks
  Change in score on HAM-D-17 item # 1 "Depressed mood" (Hieronymus et al., 2015)
Absolute change in "inflammatory depressive symptoms" | 8 weeks
  Some depression symptoms such as anhedonia, fatigue and sleep or appetite disturbances may be more strongly linked with inflammation than others (Jokela, Virtanen et al. 2016, Miller, Haroon et al. 2016). "Inflammatory depressive symptoms", will defined as defined as a total composite score of the following items from the Patient Health Questionnaire-9 (PHQ-9)) (Kroenke, Spitzer et al. 2001): item 3 (sleep problems), item 4 (lack of energy), and item 5 (appetite disturbance).
Improvement in functioning and quality of life. | 8 weeks
  WHO Disability Assessment Schedule
Absolute change in general Anxiety symptoms | 8 weeks
  Generalized Anxiety Disorder-7 (GAD-7), self rating scale
Absolute change in IL-6 and TNF-alpha | 8 weeks
  IL-6, TNF-alpha (pg/ml)
Absolute change in CRP, leptin, adiponectin | 8 weeks
  CRP, leptin, adiponectin (mg/L)
Absolute change in oxidative stress marker F2 Isoprostanes | 8 weeks
  F2-Isoprostanes (ng/ml)
Absolute change in oxidative stress marker 8-OHdG | 8 weeks
  8-OH 2-deoxyguanosine (pmol/mikrog DNA)
Absolute change in oxidative stress marker glutathione | 8 weeks
  Glutathione (mikroM)
Absolute change in metabolic markers | 8 weeks
  Cholesterol, triglycerides, glucose (mg/dL)
Absolute change in antioxidant glutathione peroxidase | 8 weeks
  Glutathione peroxidase (nmole NADPH/ml/min)
Absolute change in vascular cell adhesion molecule (VCAM) and intracellular adhesion molecule (ICAM) | 8 weeks
  ICAM, VCAM (ng/ml)
Absolute change in leukocyte telomerase activity | 8 weeks
  leukocyte telomerase activity (units/10 000 cells)
Absolute change in leukocyte telomere length | 8 weeks
  leukocyte telomere length (base pairs)
Absolute change in circulating cell-free mitochondrial DNA (ccf mtDNA) | 8 weeks
  ccf mtDNA (units/mikrolitre plasma)
Number of dropouts (due to side effects) | 8 weeks
  Number of dropouts (due to side effects)
Remission in depressive symptoms | 8 weeks
  "Remission" is defined as post-treatment HAM-D-17 ratings of < 7

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Dept of Psychiatry, Lund, Sweden

REFERENCES:
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Raison CL, Demetrashvili M, Capuron L, Miller AH. Neuropsychiatric adverse effects of interferon-alpha: recognition and management. CNS Drugs. 2005;19(2):105-23. doi: 10.2165/00023210-200519020-00002. PMID 15697325
- [Background] Jokela M, Virtanen M, Batty GD, Kivimaki M. Inflammation and Specific Symptoms of Depression. JAMA Psychiatry. 2016 Jan;73(1):87-8. doi: 10.1001/jamapsychiatry.2015.1977. No abstract available. PMID 26579988
- [Background] Raison CL, Miller AH. Is depression an inflammatory disorder? Curr Psychiatry Rep. 2011 Dec;13(6):467-75. doi: 10.1007/s11920-011-0232-0. PMID 21927805
- [Background] Miller AH, Haroon E, Felger JC. Therapeutic Implications of Brain-Immune Interactions: Treatment in Translation. Neuropsychopharmacology. 2017 Jan;42(1):334-359. doi: 10.1038/npp.2016.167. Epub 2016 Aug 24. PMID 27555382
- [Background] Rapaport MH, Nierenberg AA, Schettler PJ, Kinkead B, Cardoos A, Walker R, Mischoulon D. Inflammation as a predictive biomarker for response to omega-3 fatty acids in major depressive disorder: a proof-of-concept study. Mol Psychiatry. 2016 Jan;21(1):71-9. doi: 10.1038/mp.2015.22. Epub 2015 Mar 24. PMID 25802980
- [Background] Lindqvist D, Epel ES, Mellon SH, Penninx BW, Revesz D, Verhoeven JE, Reus VI, Lin J, Mahan L, Hough CM, Rosser R, Bersani FS, Blackburn EH, Wolkowitz OM. Psychiatric disorders and leukocyte telomere length: Underlying mechanisms linking mental illness with cellular aging. Neurosci Biobehav Rev. 2015 Aug;55:333-64. doi: 10.1016/j.neubiorev.2015.05.007. Epub 2015 May 18. PMID 25999120
- [Background] Babcock T, Helton WS, Espat NJ. Eicosapentaenoic acid (EPA): an antiinflammatory omega-3 fat with potential clinical applications. Nutrition. 2000 Nov-Dec;16(11-12):1116-8. doi: 10.1016/s0899-9007(00)00392-0. No abstract available. PMID 11118844
- [Background] Rangel-Huerta OD, Aguilera CM, Mesa MD, Gil A. Omega-3 long-chain polyunsaturated fatty acids supplementation on inflammatory biomakers: a systematic review of randomised clinical trials. Br J Nutr. 2012 Jun;107 Suppl 2:S159-70. doi: 10.1017/S0007114512001559. PMID 22591890
- [Background] Calder PC. Omega-3 polyunsaturated fatty acids and inflammatory processes: nutrition or pharmacology? Br J Clin Pharmacol. 2013 Mar;75(3):645-62. doi: 10.1111/j.1365-2125.2012.04374.x. PMID 22765297
- [Background] Kiecolt-Glaser JK, Epel ES, Belury MA, Andridge R, Lin J, Glaser R, Malarkey WB, Hwang BS, Blackburn E. Omega-3 fatty acids, oxidative stress, and leukocyte telomere length: A randomized controlled trial. Brain Behav Immun. 2013 Feb;28:16-24. doi: 10.1016/j.bbi.2012.09.004. Epub 2012 Sep 23. PMID 23010452
- [Background] Saunders EF, Ramsden CE, Sherazy MS, Gelenberg AJ, Davis JM, Rapoport SI. Omega-3 and Omega-6 Polyunsaturated Fatty Acids in Bipolar Disorder: A Review of Biomarker and Treatment Studies. J Clin Psychiatry. 2016 Oct;77(10):e1301-e1308. doi: 10.4088/JCP.15r09925. PMID 27631140
- [Background] Bloch MH, Hannestad J. Omega-3 fatty acids for the treatment of depression: systematic review and meta-analysis. Mol Psychiatry. 2012 Dec;17(12):1272-82. doi: 10.1038/mp.2011.100. Epub 2011 Sep 20. PMID 21931319
- [Background] Mocking RJ, Harmsen I, Assies J, Koeter MW, Ruhe HG, Schene AH. Meta-analysis and meta-regression of omega-3 polyunsaturated fatty acid supplementation for major depressive disorder. Transl Psychiatry. 2016 Mar 15;6(3):e756. doi: 10.1038/tp.2016.29. PMID 26978738
- [Background] Su KP, Huang SY, Chiu CC, Shen WW. Omega-3 fatty acids in major depressive disorder. A preliminary double-blind, placebo-controlled trial. Eur Neuropsychopharmacol. 2003 Aug;13(4):267-71. doi: 10.1016/s0924-977x(03)00032-4. PMID 12888186
- [Background] Hieronymus F, Emilsson JF, Nilsson S, Eriksson E. Consistent superiority of selective serotonin reuptake inhibitors over placebo in reducing depressed mood in patients with major depression. Mol Psychiatry. 2016 Apr;21(4):523-30. doi: 10.1038/mp.2015.53. Epub 2015 Apr 28. PMID 25917369
- [Derived] Suneson K, Soderberg Veiback G, Lindahl J, Tjernberg J, Stahl D, Ventorp S, Angeby F, Lundblad K, Wolkowitz OM, Lindqvist D. Omega-3 fatty acids for inflamed depression - A match/mismatch study. Brain Behav Immun. 2024 May;118:192-201. doi: 10.1016/j.bbi.2024.02.029. Epub 2024 Mar 1. PMID 38432599
- [Derived] Suneson K, Angeby F, Lindahl J, Soderberg G, Tjernberg J, Lindqvist D. Efficacy of eicosapentaenoic acid in inflammatory depression: study protocol for a match-mismatch trial. BMC Psychiatry. 2022 Dec 19;22(1):801. doi: 10.1186/s12888-022-04430-z. PMID 36536364